CLINICAL TRIAL: NCT04887389
Title: Cariostatic and Remineralizing Effects of Three Different Dental Varnishes (A Clinical Trial)
Brief Title: Cariostatic and Remineralizing Effects of Three Different Dental Varnishes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nisreen Ibrahim khan (Other)
Responsible Party: Sponsor-Investigator, Nisreen Ibrahim khan, Lecturer of Dental Public Health and Preventive Dentistry, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A07071020
Record Dates: First submitted 2021-05-05; First posted 2021-05-14 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2022-06

CONDITIONS: Dental Caries in Children; Cariostatic Agent; Resistance, Dental Caries; Fluoride Varnishes
Keywords: Dental caries prevention; NSF (nano silver fluoride); n-HAP (Nano hydroxyapatite ); NaF ( Sodium Fluoride); ICDAS II; Enamel biopsy
MeSH Terms: conditions — Dental Caries | interventions — N-Ethylmaleimide-Sensitive Proteins; Bifluorid 12

STUDY DESIGN:
Intervention Model Description: Selected children will be divided randomly into three groups:
  * Group 1: Children receiving Nano Silver Fluoride varnish (NSF) (n =39).
  * Group 2 Children receiving Nano-hydroxyapatite varnish (n = 37).
  * Group 3: Children receiving Sodium Fluoride Varnish (n = 39) Procedure for material application The application of single drop (0.1 mL) of either (5%) NSF, (10%) n-HAP, (5%) NaF varnishes with a disposable micro-applicator tip for 10 seconds. NSF will be used in a single application and no repetition. While n-HAP, NaF varnishes will be applied each 6 months .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group of • Nano Silver Fluoride varnish ( NSF) (Experimental): Selected children will be divided randomly into three groups:
  Group 1: Children receiving Nano Silver Fluoride varnish (NSF) (n =50).
  Interventions: Drug: Nano Silver Fluoride varnish
- group of Nano hydroxyapatite varnish (n-HAP) (Experimental): Group 2 Children receiving Nano-hydroxyapatite varnish (n = 50)
  Interventions: Drug: nano-hydroxyapatite varnish
- group of Sodium Fluoride Varnish (NaF) (Experimental): Group 3: Children receiving Sodium Fluoride Varnish (n = 50)
  Interventions: Drug: sodium Fluoride Varnish

INTERVENTIONS:
Drug: Nano Silver Fluoride varnish — Nano Silver Fluoride(5%) is a new experimental formulation containing silver nanoparticles, chitosan and fluoride combines preventive and antimicrobial properties. It is a yellow solution and safe to be used in humans
  Other Names: ( NSF)
  Arms: Group of • Nano Silver Fluoride varnish ( NSF)
Drug: nano-hydroxyapatite varnish — nano-hydroxyapatite (10%) has antibacterial effect, higher solubility, surface energy and bioactivity and its structure is similar to dental apatite.
  Other Names: (n-HAP)
  Arms: group of Nano hydroxyapatite varnish (n-HAP)
Drug: sodium Fluoride Varnish — Fluoride varnish (5%) applied every six months is effective in preventing caries in the primary and permanent dentition of children and adolescents
  Other Names: NaF
  Arms: group of Sodium Fluoride Varnish (NaF)

SUMMARY:
This study is a randomly, controlled, prospective in vivo study.

The objective of this study is:

To evaluate the cariostatic and re-mineralizing effects of Nano silver fluoride, Nano Hydroxyapatite and sodium fluoride varnishes in caries prevention through:

1. Clinical evaluation using international caries detection and assessment system (ICDAS II visual scoring criteria)
2. Calcium and fluoride content using enamel biopsy

DETAILED DESCRIPTION:
Dental caries is a chronic, multi factorial, transmissible, infectious disease. Caries prevalence in young children in Egypt is very high, and most of the decayed teeth are left untreated, The increase prevalence of dental caries in children globally and in developing countries such as Egypt particularly makes the need for preventive treatment is necessary, one of the ways to prevent dental caries is the application of fluoride which can prevent dental caries by inhibiting demineralization of the crystal structures inside the tooth and enhancing remineralization.

Subsequently over the years various topical fluoride agents have been evolved but NaF (a 22,600 ppm F- preparation) is the most commonly used agent, Based on systematic studies, 5% NaF varnish was more effective in re-mineralizing early enamel caries.

Another anti caries product is a nano-hydroxyapatite (n-HAP), it has antibacterial effect, higher solubility, surface energy and bio activity, there are several studies concluded that 10% (n-HAP) may be optimal for remineralization of early enamel caries Nano-Silver Fluoride (NSF) is a new experimental formulation containing silver nanoparticles, it was introduced by Targino AG et al.(2014) to combat the problem of black discoloration of Silver Diamine Fluoride. It is safe to be used in humans and has effective antimicrobial properties against the pathogens responsible for the development of dental caries.

most of the studies have been evaluated the effectiveness of anti-caries agent in In Vitro and to the best of our knowledge, there are no published studies in Egypt on the effectiveness of these agent. As such, due to the continuous development of new remineralizing agents, research is needed to investigate the newer remineralizing agents under different circumstances. The present study will be carried out to evaluate the efficacy of Nano silver fluoride, Nano Hydroxyapatite and Sodium fluoride varnishes in caries prevention.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria of participated children :

  1. Age rang 7-10 years.
  2. Teeth with score 0, 1 or 2 according to (international caries detection and assessment system) ICDAS II index.
  3. Patient did not receive any re-mineralizing agent other than the regular toothpaste during the past three months.
  4. No known history of allergy against silver particles or colophonium.
  5. written informed consent from the parents/guardians.

     Exclusion Criteria:

  <!-- -->

  1. Teeth with score 3 or more according to ICDAS II index.
  2. Partially erupted permanent teeth.

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 115 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
a. Clinical evaluation using international caries detection and assessment system (ICDAS II visual scoring criteria | 1. All children will be assessed clinically in four visits along one year, at the baseline as well as at 3rd, 6th and 12th month of follow up visit
  After taking the personal data of the participant, dental examination will be conducted by one trained and calibrated examiner under the standard situation including semi-supine position of the subject, good illumination and taking into account all methods of infection control.
  Baseline dental examination for all surfaces of included teeth according to ICDAS II was recorded. Only the surfaces with 0, 1 and 2 score will be included in the follow up assessment (Drying of the tooth surface is the key for detecting non-cavitated lesions).
  Diagnostic criteria for newly dental caries :
  In order to compare the preventive efficacy of the three preventive agent, any change in the baseline recording of score 0, 1, or 2 will be recorded in each visit of all three groups, and an comparison will be made between the mean of tooth surfaces with score 0, 1 or 2 in the baseline visit and during all follow-up visits in each group and after that comparing among all groups.
Enamel biopsy for detecting Calcium and Fluoride content . | Fluoride and calcium content will be evaluated at the baseline as well as at the last follow-up visit through study completion, an average of 1 year"
  The tooth on which the biopsy had to be done will be isolated with the help of cotton rolls and high volume suction to eliminate any chances of saliva contamination. Sticking plaster will be used to cover the tooth to be subjected for biopsy. A 6 mm circular punch will be made in the sticking plaster keeping in mind that it should be present on the buccal surface of molar. A 6 mm non-fluoride containing circular blotting paper will wetted with 5 µL of 30% phosphoric acid and immediately placed on the punched window for 4 s . This filter paper will then transferred to plastic tube which had 0.1 ml of double distilled water pipetted using a micro-pipette. Equal amount of total ionic strength adjustment buffer (TISAB-II) will added using a micropipette to the plastic tube, after which it will be stored for 3 days. After that it will send to laboratory for fluoride and calcium analysis.At the end -fluoride varnish will be applied to the surface.

CONTACTS AND LOCATIONS:
Overall Officials: Salwa A Hegazy, PhD, Principal Investigator — Head of Dental Public Health department
Locations (1):
- Faculty of Dentistry / Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abbass MMS, Mahmoud SA, El Moshy S, Rady D, AbuBakr N, Radwan IA, Ahmed A, Abdou A, Al Jawaldeh A. The prevalence of dental caries among Egyptian children and adolescences and its association with age, socioeconomic status, dietary habits and other risk factors. A cross-sectional study. F1000Res. 2019 Jan 3;8:8. doi: 10.12688/f1000research.17047.1. eCollection 2019. PMID 30854195
- [Result] Azarpazhooh A, Main PA. Fluoride varnish in the prevention of dental caries in children and adolescents: a systematic review. Tex Dent J. 2008 Apr;125(4):318-37. No abstract available. PMID 18491761
- [Result] Chu CH, Mei ML, Lo EC. Use of fluorides in dental caries management. Gen Dent. 2010 Jan-Feb;58(1):37-43; quiz 44-5, 79-80. PMID 20129891
- [Result] Huang SB, Gao SS, Yu HY. Effect of nano-hydroxyapatite concentration on remineralization of initial enamel lesion in vitro. Biomed Mater. 2009 Jun;4(3):034104. doi: 10.1088/1748-6041/4/3/034104. Epub 2009 Jun 5. PMID 19498220
- [Result] Pepla E, Besharat LK, Palaia G, Tenore G, Migliau G. Nano-hydroxyapatite and its applications in preventive, restorative and regenerative dentistry: a review of literature. Ann Stomatol (Roma). 2014 Nov 20;5(3):108-14. eCollection 2014 Jul. PMID 25506416
- [Result] Targino AG, Flores MA, dos Santos Junior VE, de Godoy Bene Bezerra F, de Luna Freire H, Galembeck A, Rosenblatt A. An innovative approach to treating dental decay in children. A new anti-caries agent. J Mater Sci Mater Med. 2014 Aug;25(8):2041-7. doi: 10.1007/s10856-014-5221-5. Epub 2014 May 13. PMID 24818873